CLINICAL TRIAL: NCT02479035
Title: Red Raspberries and Insulin Action: Understanding the Role of Red Raspberry Consumption on Oxidative Stress- and Inflammatory- Mediated Insulin Action in Humans
Brief Title: Red Raspberries on Insulin Action and Oxidative Stress
Acronym: RRB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Nutrition Research Center, Illinois Institute of Technology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: IRB2015-030
Record Dates: First submitted 2015-06-19; First posted 2015-06-23 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-08

CONDITIONS: Insulin Resistant
Keywords: insulin sensitive; insulin resistant; red raspberry; polyphenols; bioavailability

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Red raspberry meal 1 (Active Comparator): ~125 g fresh weight (1 cup equivalent)
  Interventions: Dietary Supplement: Red raspberry meal 1
- Red raspberry meal 2 (Active Comparator): ~250 g fresh weight (2 cup equivalent)
  Interventions: Dietary Supplement: Red raspberry meal 2
- Control meal (Placebo Comparator): 0 g red raspberry
  Interventions: Dietary Supplement: Control meal

INTERVENTIONS:
Dietary Supplement: Red raspberry meal 1 — ~125 g fresh weight (1 cup equivalent)
  Arms: Red raspberry meal 1
Dietary Supplement: Red raspberry meal 2 — ~250 g fresh weight (2 cup equivalent)
  Arms: Red raspberry meal 2
Dietary Supplement: Control meal — 0 g red raspberry
  Arms: Control meal

SUMMARY:
The purpose of this study is to investigate the relative bioavailability and absorption/kinetic profile of red raspberry polyphenols consumed with a meal and further to determine the relationship of these findings on meal-associated metabolic- oxidative- and inflammatory- responses in relatively insulin sensitive and insulin resistant individuals.

DETAILED DESCRIPTION:
The proposed study is a randomized, 3-arm, diet-controlled, cross-over study using a multi-sampling postprandial paradigm to evaluate the relative bioavailability and absorption/kinetic profile of red raspberry polyphenols consumed with a typical American breakfast meal and further to determine the relationship of these findings on meal-associated metabolic- oxidative- and inflammatory- responses in relatively insulin sensitive and insulin resistant individuals. A planned sample size of 24 will be recruited into the study. This study will require one initial screening visit, 1 pre-study visit, and 3 study visits. This study will take 4-6 weeks per subject to complete.

The trial will initiate with a screening visit, which will last for about 1-1.5 hours and include measuring subjects' height, weight, waist circumference, fasting blood glucose, insulin sensitivity, body temperature, blood pressure and heart rate as well as collecting general eating, health and exercise habits via questionnaire.

If willing and eligible to participate, a 3-day food record (2 weekdays and 1 weekend) will be given to be completed over the following week to assess subject's baseline dietary intake patterns. Information will be used to help subjects adopt a relatively low polyphenolic diet over the course of the study. Prior to each postprandial study visit, a dinner meal will be provided the day before the study visit to help control for visit to visit variability in due to differences in meals the night before the study visit.

Subjects will arrive at the center in a fasting state for at least 10 hours, well hydrated and rested (with normal sleep). Each study visit will require blood draws throughout the visit. After evaluation of subject's health status (via anthropometric, vital sign and blood glucose measurements and in-person interview), a qualified health professional will place a catheter in subject's arm for the purpose of multiple blood sample collections and take the initial blood draw in the fasting state. Each subject will be randomized to receive 1 of 3 meal treatments: Control meal (0 g red raspberry), red raspberry meal 1 [~125 g fresh weight (1 cup equivalent)] or red raspberry meal 2 [~250 g fresh weight (2 cup equivalent)], based on randomization sequence on 3 Study Day Visits. At each Study visit, after the first blood draw (0 h), subjects will be served with the standard breakfast meal (a moderate to high fat/carbohydrate) along with fruit variable based on the order randomly selected by computer generated sequence. From this point forward, blood collection will occur at the following time points: 0.5 h, 1 h, 2 h, 3 h, 4 h, 5 h, 6 h, 6.5 h, 7 h, 8 h and 24 h to test for polyphenol metabolites and other metabolic markers. After the 6h blood draw, a standardized lunch meal (polyphenol free) will be provided to subjects. After the 8 h blood draw, the catheter will be removed from subjects arm. Subject will be provided with a dinner meal (low polyphenol) to take home and asked not to consume anything else other than the provided dinner meal except plain water. Subject will be scheduled to come back the next morning for the 24 h blood sample collection.

ELIGIBILITY:
Inclusion Criteria:

* Fasting blood sugar between 100-125 mg/dL and fasting insulin concentration ≥ 8 uIU/mL for Prediabetes,insulin-resistant group
* Fasting blood sugar < 100 mg/dL and the homeostasis model assessment method of insulin resistance (HOMA-IR) (glucose [in millimoles per liter] × insulin [in microunits per milliliter]/22.5) values less than 1 for reference/control group.
* Aged between 20 to 60 years old male/female
* Non-smoker or Past smokers: abstinence for less than 2 years
* No clinical evidence of cardiovascular, metabolic, respiratory, renal, gastrointestinal or hepatic disease
* Not taking any medications or dietary supplements that would interfere with outcomes of the study.

Exclusion Criteria:

* Men and women who smoke
* Men and women with known or suspected food intolerance, allergies or hypersensitivity to the study materials or closely related compound or any their stated ingredients.
* Men and women known to have/diagnosed with diabetes mellitus
* Men and women who have fasting blood glucose concentrations ≥126 mg/dL
* Men and women with documented vascular disease, e.g., heart failure, myocardial infarction, stroke, angina, related surgeries.
* Men and women with cancer other than non-melanoma skin cancer in previous 5 years.
* interfere with the outcomes of the study; e.g., antioxidant supplements, anti-inflammation, lipid lowering medication. Subjects may choose to go off dietary supplements (requires 30 days washout).
* Men and women who have donated blood within 3 months of the screening visit and blood donors/participants for whom participation in this study will result in having donated more than 1500 milliliters of blood in the previous 12 months.
* Substance (alcohol or drug) abuse within the last 2 years.
* Excessive coffee and tea consumers (> 4 cups/day)
* Unstable weight: gained or lost weight +/- 5 lbs in previous 3 months
* Women who are known to be pregnant or who are intending to become pregnant over the course of the study and women who are lactating

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-06-15 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
Changes in plasma metabolic markers over 8 h after consuming iso-caloric meals prepared with and without red raspberry | 8 hours
  The influence of red raspberry consumption on metabolic markers (insulin and glucose)

SECONDARY OUTCOMES:
Characterization of plasma polyphenol metabolites and concentration differences over 8 after consuming iso-caloric meals with and without red raspberry | 8 hours
  plasma polyphenol metabolites concentration
Changes in fasting plasma metabolites over 24 h after consuming iso-caloric meals prepared with and without red raspberry | 24 hr
  Comparing fasting baseline plasma metabolic markers to 24 hr fasting plasma metabolites after consuming iso-caloric meals prepared with and without red raspberry
Changes in fasting plasma metabolic markers over 24 h after consuming iso-caloric meals prepared with and without red raspberry | 24 hr
  Comparing fasting baseline plasma metabolic markers to 24 hr fasting plasma metabolic markers after consuming iso-caloric meals prepared with and without red raspberry

OTHER OUTCOMES:
Changes in inflammation and oxidative markers over 8 after consuming iso-caloric meals prepared with and without red raspberry | 8 hours
  The influence of red raspberry consumption on inflammation and oxidative markers

CONTACTS AND LOCATIONS:
Overall Officials: Britt Burton-Freeman, Ph.D, Principal Investigator — Illinois Institute of Technology
Locations (1):
- Clinical Nutrition Research Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao D, Zhu L, Edirisinghe I, Fareed J, Brailovsky Y, Burton-Freeman B. Attenuation of Postmeal Metabolic Indices with Red Raspberries in Individuals at Risk for Diabetes: A Randomized Controlled Trial. Obesity (Silver Spring). 2019 Apr;27(4):542-550. doi: 10.1002/oby.22406. Epub 2019 Feb 14. PMID 30767409